## TITLE:

Effectiveness of nasal suction in infants with bronchiolitis using a NoseFrida vs. bulb syringe: a prospective observational study

NCT 04599101

Date: 01/04/2024

Statistical Analysis Plan

## Statistical Analysis Plan

Effectiveness of nasal suction in infants with bronchiolitis using a NoseFrida vs. bulb syringe: a prospective observational study

v. 1.0 04 Jan 2024

Demographic and outcome data will be stratified by study arm and summarized using mean (SD) or median (IQR) for continuous data and compared using a t-test or Mann-Whitney U test. Categorical data will be summarized using median and full range and compared using Fisher's exact test